CLINICAL TRIAL: NCT00803790
Title: A 2-Part, Open-Label, Randomized, Crossover Study to Evaluate the Bioequivalence of the 70-mg Alendronate/5600 IU Vitamin D3 Final Market Combination Tablet to a 70-mg Alendronate Marketed Tablet, and the Relative Bioavailability of Vitamin D3
Brief Title: A Study of the Bioequivalence of 70-mg Alendronate and 70-mg Alendronate in Combination With 5600 IU Vitamin D (MK0217A-253)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0217A-253; 2008_595
Record Dates: First submitted 2008-12-04; First posted 2008-12-08 (Estimated); Results first posted 2011-05-09 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

ARMS (4):
- Sequence 1- alendronate+vitamin D combination then alendronate (Experimental): Participants in Part 1 received 70mg alendronate+5600 International Units (IU) vitamin D combination tablet in Period 1 followed by 70mg alendronate tablet in Period 2. A washout of at least 12 days separated each treatment period.
  Interventions: Drug: alendronate sodium+vitamin D combination; Drug: Comparator: alendronate
- Sequence 2 alendronate then alendronate+vitamin D combination (Experimental): Participants in Part 1 received 70mg alendronate tablet in Period 1 followed by 70mg alendronate+5600 IU vitamin D combination tablet in Period 2. A washout of at least 12 days separated each treatment period.
  Interventions: Drug: alendronate sodium+vitamin D combination; Drug: Comparator: alendronate
- Sequence 3 alendronate+vitamin D combination then vitamin D (Experimental): Participants in Part 2 received 70mg alendronate+5600 IU vitamin D combination tablet in Period 1 followed by a single dose of 5600 IU vitamin D, administered as two 2800 IU tablets in Period 2. A washout of at least 12 days separated each treatment period.
  Interventions: Drug: alendronate sodium+vitamin D combination; Dietary Supplement: Comparator: Vitamin D
- Sequence 4- vitamin D then alendronate+vitamin D combination (Experimental): Participants in Part 2 received a single dose of 5600 IU vitamin D, administered as two 2800 IU tablets in Period 1 followed by a 70mg alendronate+5600 IU vitamin D combination tablet in Period 2. A washout of at least 12 days separated each treatment period.
  Interventions: Drug: alendronate sodium+vitamin D combination; Dietary Supplement: Comparator: Vitamin D

INTERVENTIONS:
Drug: alendronate sodium+vitamin D combination — A single dose tablet of 70mg alendronate sodium+5600 IU vitamin D combination tablet in one treatment period of each sequence.
Drug: Comparator: alendronate — A single dose tablet of 70mg alendronate in one treatment period of each sequence.
  Arms: Sequence 1- alendronate+vitamin D combination then alendronate; Sequence 2 alendronate then alendronate+vitamin D combination
Dietary Supplement: Comparator: Vitamin D — Two tablets of 2800 IU vitamin D, totaling 5600 IU, in one treatment period of each sequence.
  Arms: Sequence 3 alendronate+vitamin D combination then vitamin D; Sequence 4- vitamin D then alendronate+vitamin D combination

SUMMARY:
This study will evaluate the bioequivalence of alendronate in combination with vitamin D compared to alendronate alone and the bioequivalence of vitamin D in combination with alendronate compared to vitamin D alone.

This was an open-label, randomized, 2-part, crossover study. Each participant participated in one part of the study only (i.e., each participant participated only in Part I or only in Part II). Participants entered the study sequentially within each part of the study. A washout of at least 12 days separated each treatment period within each part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or nonpregnant female age 18 to 85 years
* female of childbearing potential on appropriate method of contraception and not nursing
* Body Mass Index (BMI) less than or equal to 30 kg/m2
* subject is in good health

Exclusion Criteria:

* mental or legal incapacitation
* received bisphosphonate treatment within 3 months of enrollment.
* unable to sit or stand upright for at least 2 hours
* unwilling to refrain from consumption of alcohol or caffeinated products from 24 hours prior and 36 hours after study drug administration
* unwilling to limit alcohol consumption to no more than 2 drinks per day
* unwilling to limit caffeinated products to the equivalent of 4 cups of coffee per day or equivalent.
* unwilling to refrain from smoking during the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2006-05; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Denker AE, Lazarus N, Porras A, Ramakrishnan R, Constanzer M, Scott BB, Chavez-Eng C, Woolf E, Maganti L, Larson P, Gottesdiener K, Wagner JA. Bioavailability of alendronate and vitamin D(3) in an alendronate/vitamin D(3) combination tablet. J Clin Pharmacol. 2011 Oct;51(10):1439-48. doi: 10.1177/0091270010382010. Epub 2010 Dec 8. PMID 21148044

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a randomized, 2-part, crossover study. Each participant participated in one part of the study only (i.e., each participant participated only in Part I or only in Part II). A washout of at least 12 days separated each treatment period within each part of the study. 318 participants were enrolled (251 in Part 1 and 67 in Part 2).
Groups:
- Part 1 Alendronate+Vitamin D Combo, Then Alendronate: Participants in Part 1 received a single dose of 70mg alendronate+5600 International Units (IU) vitamin D combination tablet in Period 1 followed by a single dose of 70mg alendronate tablet in Period 2. A washout of at least 12 days separated each treatment period.
- Part 1 Alendronate, Then Alendronate+Vitamin D Combo: Participants in Part 1 received a single dose of 70mg alendronate tablet in Period 1 followed by a single dose of 70mg alendronate+5600 IU vitamin D combination tablet in Period 2. A washout of at least 12 days separated each treatment period.
- Part 2 Alendronate+Vitamin D Combo, Then Vitamin D: Participants in Part 2 received a single dose of 70mg alendronate+5600 IU vitamin D combination tablet in Period 1 followed by a single dose of 5600 IU vitamin D, administered as two 2800 IU tablets in Period 2. A washout of at least 12 days separated each treatment period.
- Part 2 Vitamin D, Then Alendronate+Vitamin D Combo: Participants in Part 2 received a single dose of 5600 IU vitamin D, administered as two 2800 IU tablets in Period 1 followed by a single dose of 70mg alendronate+5600 IU vitamin D combination tablet in Period 2. A washout of at least 12 days separated each treatment period.
Period: Period 1
Arm/Group | Part 1 Alendronate+Vitamin D Combo, Then Alendronate | Part 1 Alendronate, Then Alendronate+Vitamin D Combo | Part 2 Alendronate+Vitamin D Combo, Then Vitamin D | Part 2 Vitamin D, Then Alendronate+Vitamin D Combo
Started | 125 | 126 | 32 | 35
Completed | 116 | 114 | 31 | 31
Not Completed | 9 | 12 | 1 | 4
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 6 | 0 | 0
Not completed — positive drug screen or personal reasons | 0 | 3 | 0 | 4
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Period: Period 2
Arm/Group | Part 1 Alendronate+Vitamin D Combo, Then Alendronate | Part 1 Alendronate, Then Alendronate+Vitamin D Combo | Part 2 Alendronate+Vitamin D Combo, Then Vitamin D | Part 2 Vitamin D, Then Alendronate+Vitamin D Combo
Started | 116 | 114 | 31 | 31
Completed | 114 | 114 | 30 | 30
Not Completed | 2 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Positive Drug Screen or Personal Reasons | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 1: Alendronate+vitamin D combo, then alendronate: In Period 1 participants received a single dose of 70mg alendronate+5600 IU vitamin D combination tablet, and in Period 2 a single dose of 70mg alendronate tablet. A washout of at least 12 days separated each treatment period.
  Alendronate, then alendronate+vitamin D combo: In Period 1 participants received 70mg alendronate tablet, and in Period 2 a single dose of 70mg alendronate+5600 IU vitamin D combination tablet. A washout of at least 12 days separated each treatment period.
- Part 2: Alendronate+vitamin D combo, then vitamin D: In Period 1 participants received a single dose of 70mg alendronate+5600 IU vitamin D combination tablet, and in Period 2 a single dose of 5600 IU vitamin D, administered as 2 x 2800 IU tablets. A washout of at least 12 days separated each treatment period.
  Vitamin D, then alendronate+vitamin D combo: In Period 1 participants received a single dose of 5600 IU vitamin D, administered as 2 x 2800 IU tablets, and in Period 2 a single dose of 70mg alendronate+5600 IU vitamin D combination tablet. A washout of at least 12 days separated each treatment period.
- Total: Total of all reporting groups
Arm/Group | Part 1 | Part 2 | Total
Number analyzed (Participants) | 251 | 67 | 318
Age, Customized [Number; unit: participants]
  Between 18 and 78 years | 251 | 67 | 318
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 29 | 161
  Male | 119 | 38 | 157

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Urinary Excretion of Alendronate
Description: Bioequivalence was demonstrated by measuring the total urinary excretion of alendronate which was determined over a 36-hour period following single dose administration of 70-mg alendronate+5600 International Units (IU) vitamin D combination tablet and 70mg alendronate tablet alone. Urine for each treatment period was collected at -2 to 0 hours predose, 0 to 8, 8 to 24, and 24 to 36 hours postdose on Days 1 and 2.
Time Frame: Day 1-2 across the 36 hour urinary collection period (Periods 1 and 2)
Population: 220 participants of the 251 enrolled in Part 1 were included in the statistical analysis. 31 participants were excluded: 23 were enrolled but did not complete both study periods and 8 participants had incomplete urine profiles in one or both periods.
Measure: Least Squares Mean (Standard Deviation); unit: μg
Groups:
- Alendronate+Vitamin D Combo: Single dose of 70mg alendronate+5600 IU vitamin D combination tablet
- Alendronate: Single dose of 70mg alendronate tablet
Arm/Group | Alendronate+Vitamin D Combo | Alendronate
Number analyzed (Participants) | 220 | 220
μg | 133.6 (189.2) | 132.2 (273.4)
Statistical Analysis 1: Comparison: Alendronate+Vitamin D Combo vs Alendronate; Test type: Superiority or Other; least square mean ratio = 1.01, 90% CI 2-sided [0.92 to 1.11]

2. Primary Outcome: Part II: AUC (Area Under the Plasma Concentration-time Curve) of Vitamin D
Description: The serum vitamin D pharmacokinetic parameter was calculated following the treatment of 70mg alendronate+5600 IU vitamin D combination tablet and 5600 IU vitamin D tablet on Day 1: area under the plasma concentration-time curve (AUC0-80hr). Serum samples for determination of vitamin D concentrations were obtained at -2 and 0 hrs predose on Day 1 and at 2, 3, 5, 7, 9, 12, 16, 24, 36, 48, 72 and 80 hours post dose for each treatment period.
Time Frame: Day 1 across the 80-hour plasma collection period (Period 1 and 2)
Population: 60 participants of the 67 enrolled in Part 2 were included in the statistical analysis. 7 participants that were enrolled, but did not complete both study periods were excluded.
Measure: Least Squares Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Alendronate+Vitamin D Combo: A single dose of 70mg alendronate+5600 IU vitamin D combination tablet
- Vitamin D: Single dose of 5600 IU vitamin D administered as 2 x 2800 IU tablets
Arm/Group | Alendronate+Vitamin D Combo | Vitamin D
Number analyzed (Participants) | 60 | 60
ng*hr/mL | 490.2 (259.6) | 518.7 (269.8)
Statistical Analysis 1: Comparison: Alendronate+Vitamin D Combo vs Vitamin D; Least squares mean ratio for AUC 0-80 hr for vitamin D following administration of combination tablet and vitamin D alone. No correction for endogenous Vitamin D concentration pre-treatment was made in the analysis; Test type: Superiority or Other; Least Square Mean Ratio = 0.94, 90% CI 2-sided [0.89 to 1.00]

3. Secondary Outcome: Part II : Maximum Concentration (Cmax) of Vitamin D
Description: Serum vitamin D pharmacokinetic parameter was calculated for the following: maximum concentration of drug observed in serum (Cmax). Serum samples for determination of vitamin D concentrations were obtained at -2 and 0 hrs predose on Day 1 and at 2, 3, 5, 7, 9, 12, 16, 24, 36, 48, 72 and 80 hours post dose for each treatment period.
Time Frame: Day 1 across the 80-hour plasma collection period (Periods 1 and 2)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Deviation); unit: ng/ml
Groups:
- Alendronate+Vitamin D Combo: Single dose of 70 mg alendronate+5600 IU vitamin D combination tablet
- Vitamin D: Single dose of 5600 IU vitamin D, administered as 2 x 2800 IU tablets
Arm/Group | Alendronate+Vitamin D Combo | Vitamin D
Number analyzed (Participants) | 60 | 60
ng/ml | 12.2 (5.6) | 13.0 (5.9)
Statistical Analysis 1: Comparison: Alendronate+Vitamin D Combo vs Vitamin D; Least squares mean ratio for Cmax for vitamin D following administration of combination tablet and vitamin D alone. No correction for endogenous Vitamin D concentration pre-treatment was made in the analysis; Test type: Superiority or Other; Least Square Mean Ratio = 0.94, 90% CI 2-sided [0.88 to 1.00]

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: There were 28 missing participants whose discontinuation did not allow for them to receive the treatments assigned in both Periods 1 and 2 (Alendronate= 10, Alendronate+Vitamin D Combo= 16, Vitamin D= 2).
Arm/Group | Alendronate+Vitamin D Combo | Alendronate | Vitamin D
Serious Adverse Events (participants affected / at risk) | 0/302 | 0/241 | 0/65
Other Adverse Events (participants affected / at risk) | 21/302 | 12/241 | 9/65
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alendronate+Vitamin D Combo (N=302) | Alendronate (N=241) | Vitamin D (N=65)
Headache (Nervous system disorders) | 21 | 12 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication timelines.